CLINICAL TRIAL: NCT02391350
Title: Management Strategies for Patients With Low Back Pain and Sciatica
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Julie Fritz, Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R18HS022641 (AHRQ)
Record Dates: First submitted 2015-01-12; First posted 2015-03-18 (Estimated); Results first posted 2020-12-24 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-12

CONDITIONS: Low Back Pain; Sciatica; Physical Therapy
MeSH Terms: conditions — Low Back Pain; Sciatica | interventions — Educational Status; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Active Comparator): Patients will be managed by primary care provider with a stepped care approach supported by current practice guidelines. Initial management will include education and re-assurance for the first 4 weeks following the primary care visit. Patients in will be recommended to follow-up with their primary care provider if unsatisfied with their progress after 4 weeks. At that time decisions on further treatments and/or referrals will be made by the primary care provider in consultation with the patient consistent with usual care.
  Interventions: Behavioral: Education and re-assurance
- Early Intervention (Experimental): Patients will receive education and re-assurance in the same manner as the usual care group and will receive physical therapy during the initial 4 weeks following enrollment. Physical therapy will be based on evidence and prior research evaluating a centralizing treatment program for patients with LBP and sciatica. The first physical therapy session will be scheduled within 3 days after enrollment and 6-8 sessions will be administered in the first 4 weeks. Each session will include a brief assessment, treatment with centralizing exercises and spinal mobilizations. Mechanical traction is an optional component. Patients will be provided handouts and instructed to perform assigned exercises at home every 4-5 hours on days between sessions.
  Interventions: Behavioral: Education and re-assurance; Procedure: Physical Therapy

INTERVENTIONS:
Behavioral: Education and re-assurance — Patients are provided the Back Book and the contents are reviewed emphasizing the favorable natural history of back pain and sciatica and the importance of remaining active.
Procedure: Physical Therapy — Physical therapy will consist of repeated exercises, spinal mobilization and mechanical traction in an effort to maximize centralization of symptoms.
  Arms: Early Intervention

SUMMARY:
Low back pain and sciatica is a common condition resulting in high costs and disability for society and affected individuals. Presently there is a lack of evidence for what treatments may help this condition early in the course of care. Improved early management could reduce risks for persistent disability and high costs. The goal of this project is to examine the clinical outcomes and costs associated with adding a physical therapy program to early management of patients with low back pain and sciatica within primary care.

DETAILED DESCRIPTION:
Low back pain (LBP) is a common and costly condition. When accompanied by sciatica, risks for persistent disability and future invasive treatments increase. Most patients with LBP and sciatica enter the healthcare system in primary care. Optimal primary care management is currently unclear and little data are available to assist clinicians and inform patients of the likely effects of common options. Practice guidelines agree that imaging, spinal injections and surgeries should be reserved for patients whose symptoms do not diminish within 4-8 weeks, yet utilization rates for these procedures are increasing rapidly, partly due to the uncertainty of what options may be offered to patients for initial treatment. Physical therapy is considered an option in the initial management period, but is used inconsistently. It is currently unclear what can be expected from early physical therapy for patients with LBP and sciatica, and what if any long-term effect it may have on clinical outcomes or future healthcare utilization. The investigators research team has conducted a series of clinical trials to clarify the evidence for the most effective physical therapy procedures for patients with LBP and sciatica, and is now in a position to evaluate if the use of early, evidence-based physical therapy can reduce the risk of future disability, healthcare utilization and costs. The proposed study is a randomized trial comparing the effectiveness of usual, guideline-based initial management of newly consulting patients with LBP with sciatica with or without the addition of early physical therapy. Specific aims are to compare the clinical effectiveness, costs (direct and indirect), and cost-effectiveness of the addition of physical therapy. All patients will be managed with advice, education and medication. One group will also receive 6-8 sessions of physical therapy Outcomes will include measures of disability, pain, psychological distress, healthcare, utilization, and costs over 1 year. This study will permit an examination of the effectiveness and costs associated with the use of early physical therapy within primary care for patients with acute LBP and sciatica. The results of this study will provide needed information to assist clinicians and inform patients of their options for initial management of this common condition.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms of pain and/or numbness between the 12th rib and buttocks, which, in the opinion of the primary care provider, are originating from tissues of the lumbar region.
2. Symptoms of pain and/or numbness primarily into one leg that have extended below the knee in the last 72 hours, and correspond to a lower lumbar nerve root distribution (L4, L5, S1)
3. Current symptoms present for 90 days or fewer
4. Oswestry disability score > 20%
5. One or more of the following symptoms:

   * Positive ipsilateral or contralateral straight leg raise test (reproduction of symptoms at <70 degrees)
   * Reflex, sensory, or strength deficits in a pattern consistent with lower lumbar nerve root

Exclusion Criteria:

1. Any prior spine fusion surgery, or any surgery to the lumbosacral spine in the past year
2. Current pregnancy
3. Currently receiving treatment for LBP from another healthcare provider (e.g., chiropractic, massage therapy, injections, etc.) or any treatment for LBP in prior 6 months.
4. Judgment of primary care provider of "red flags" of a potentially serious condition including cauda equina, major or rapidly progressing neurologic deficit, fracture, cancer, infection or systemic disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2015-02; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Utah Healthcare System, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Fritz JM, Lane E, McFadden M, Brennan G, Magel JS, Thackeray A, Minick K, Meier W, Greene T. Physical Therapy Referral From Primary Care for Acute Back Pain With Sciatica : A Randomized Controlled Trial. Ann Intern Med. 2021 Jan;174(1):8-17. doi: 10.7326/M20-4187. Epub 2020 Oct 6. PMID 33017565

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from February 2015 through October, 2018. Recruitment was done in 2 health systems (University of Utah and Intermountain Healthcare) in Salt Lake City, Utah. Potential participants were identified using electronic health records and were sent a letter about the study after completing a primary care visit. A research team made follow-up telephone calls to identify those interested in meeting with a research assistant to determine eligibility and provide consent.
Period: Overall Study
Arm/Group | Usual Care | Early Intervention
Started | 110 | 110
4-week Follow-up | 106 | 105
6-month Follow-up | 100 | 96
Completed (One-year follow-up) | 98 | 93
Not Completed | 12 | 17

BASELINE CHARACTERISTICS:
Population: Missing baseline scores; sex (n = 1 EPT), age (n = 1 UC), duration of symptoms (n = 1 UC), Numeric Pain Rating Scale-leg pain intensity (n = 1 EPT), Pain Catastrophizing Scale (n = 3 EPT, n = 2 UC), Fear-Avoidance Beliefs Questionnaire physical activity subscale (n = 1 UC) and work subscale (n = 4 EPT, n = 1 UC), and EQ-5D overall health rating (n = 6 EPT, n = 3 UC).
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Early Intervention | Total
Number analyzed (Participants) | 110 | 110 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age was missing for one participant in the usual care group.
  years
    number analyzed (Participants) | 109 | 110 | 219
    (all) | 37.9 (11.2) | 40.0 (11.2) | 39.0 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender missing for one participant in Early Intervention
  Participants
    number analyzed (Participants) | 110 | 109 | 219
    Female | 59 | 48 | 107
    Male | 51 | 61 | 112
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 14 | 30
  Not Hispanic or Latino | 84 | 81 | 165
  Unknown or Not Reported | 10 | 15 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 5 | 7
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 3 | 1 | 4
  White | 89 | 92 | 181
  More than one race | 7 | 7 | 14
  Unknown or Not Reported | 3 | 2 | 5
Duration of Symptoms [Mean (Standard Deviation); unit: days] — Population: Duration of symptoms data was missing for one participant in Usual Care at Baseline
  days
    number analyzed (Participants) | 109 | 110 | 219
    (all) | 35.9 (26.8) | 35.8 (25.6) | 35.8 (26.1)
StartBack Risk Category [Count of Participants; unit: Participants] — The StartBack Risk Category describes the participant's risk for developing persistent low back pain based on physical and psychological factors. Risk stratification is based on participants' responses to 9 items about their physical and psychological symptom responses.
  Participants
    High Risk | 28 | 26 | 54
    Medium Risk | 63 | 68 | 131
    Low Risk | 19 | 16 | 35
Oswestry Disability Index [Mean (Standard Deviation); unit: units on a scale] — Measure of back pain-related disability. Scores range from 0-100 with higher scores indicating more disability due to low back pain.
  units on a scale | 35.8 (15.8) | 38.9 (13.8) | 37.3 (14.9)
Back Pain Intensity Rating [Mean (Standard Deviation); unit: units on a 0-10 scale] — Participant reported back pain intensity of 0-10 scale with higher numbers indicating greater pain intensity.
  units on a 0-10 scale | 4.8 (1.9) | 5.1 (1.8) | 5.0 (1.9)
Leg Pain Intensity Rating [Mean (Standard Deviation); unit: units on a 0-10 scale] — Participant reported intensity of pain in the leg(s) on a 0-10 scale with higher numbers indicating greater pain intensity. Population: Leg pain intensity rating was missing at baseline for one participant in the Early Intervention group.
  units on a 0-10 scale
    number analyzed (Participants) | 110 | 109 | 219
    (all) | 3.8 (2.2) | 4.3 (2.2) | 4.1 (2.2)
Euroqol 5 Dimensions (EQ-5D) [Mean (Standard Deviation); unit: units on a scale] — Participant reported measure of overall quality of life reported on five dimensions (mobility, self-care, depression/anxiety, pain/discomfort, usual activities). Scores range from 0 - 1.0 with higher scores indicating higher level of quality of life. Population: Baseline values were missing for 3 participants in Usual Care and 6 participants in Early Physical Therapy group.
  units on a scale
    number analyzed (Participants) | 107 | 104 | 211
    (all) | 0.64 (0.20) | 0.64 (0.20) | 0.64 (0.20)
Pain Catastrophizing Scale [Mean (Standard Deviation); unit: units on a scale] — Participant-reported measure of the tendency to magnify the threat value of pain. Scores range from 13-52 with higher scores indicating a higher level of pain catastrophizing. Population: Pain Catastrophizing Scale was missing at baseline for 2 participants in Usual Care and 3 participants in Early Physical Therapy group.
  units on a scale
    number analyzed (Participants) | 108 | 107 | 215
    (all) | 19.0 (11.9) | 20.9 (12.6) | 19.9 (12.3)
Fear-Avoidance Beliefs - Physical Activity [Mean (Standard Deviation); unit: units on a scale] — Participant reported measure of fear that physical activity will harm the back and should be avoided. Scores range from 0-24. Higher scores indicate greater levels of fear about physical activity. Population: Fear avoidance beliefs about physical activity data was missing for one participant in usual care group
  units on a scale
    number analyzed (Participants) | 109 | 110 | 219
    (all) | 14.0 (5.9) | 15.2 (5.7) | 14.6 (5.8)
Fear-Avoidance Beliefs - Work [Mean (Standard Deviation); unit: units on a scale] — Participant reported measure of fear that work-related activities will harm the back and should be avoided. Scores range from 0-42. Higher scores indicate greater levels of fear about work-related activities. Population: The Fear Avoidance Beliefs about Work questionnaire was missing for 4 participants in the Early Intervention group and 1 participant in the Usual Care group.
  units on a scale
    number analyzed (Participants) | 109 | 106 | 215
    (all) | 13.9 (11.8) | 15.4 (12.3) | 14.6 (12.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Oswestry Disability Index
Description: Patient-reported disability due to low back pain. Scores range from 0-100 with higher scores indicating greater disability.
Time Frame: Baseline, 4 weeks, 6 months, 1 year
Population: Missing data across follow-up is outlined by group
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | Early Intervention
Number analyzed (Participants) | 106 | 105
units on a scale
  4 Weeks | -8.8 [-11.5 to -6.0] | -17.0 [-19.7 to -14.2]
  6 months: number analyzed (Participants) | 100 | 96
  6 months | -17.0 [-19.9 to -14.2] | -22.4 [-25.3 to -19.6]
  1 year: number analyzed (Participants) | 98 | 93
  1 year | -17.7 [-20.6 to -14.8] | -22.5 [-25.4 to -19.5]

2. Secondary Outcome: Change From Baseline in Numeric Pain Ratings
Description: Separate rating for low back pain and leg pain intensity on a 0-10 scale. Higher numbers indicate greater pain intensity.
Time Frame: Baseline, 4 weeks, 6 months, 1 year
Population: Missing data reflected across follow-up points
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | Early Intervention
Number analyzed (Participants) | 106 | 105
units on a scale
  Back pain intensity 4 weeks | -1.0 [-1.4 to -0.60] | -2.4 [-2.8 to -2.1]
  Back pain intensity 6 months: number analyzed (Participants) | 100 | 96
  Back pain intensity 6 months | -1.5 [-1.9 to -1.1] | -2.3 [-2.7 to -1.9]
  Back pain intensity 1 year: number analyzed (Participants) | 98 | 93
  Back pain intensity 1 year | -1.6 [-2.0 to -1.2] | -2.6 [-3.0 to -2.2]
  Leg pain intensity 4 weeks | -1.0 [-1.4 to -0.6] | -1.8 [-2.3 to -1.4]
  Leg pain intensity 6 months: number analyzed (Participants) | 100 | 96
  Leg pain intensity 6 months | -1.9 [-2.3 to -1.5] | -1.8 [-2.2 to -1.3]
  Leg pain intensity 1 year: number analyzed (Participants) | 98 | 93
  Leg pain intensity 1 year | -1.8 [-2.2 to -1.3] | -2.2 [-2.7 to -1.8]

3. Secondary Outcome: Change From Baseline in EQ-5D
Description: Self-report measure of Quality of Life. Scores range from 0 - 1.0, with higher scores indicating greater quality of life.
Time Frame: Baseline, 4 weeks, 6 months, 1 year
Population: Missing data noted across all follow-up points
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Usual Care | Early Intervention
Number analyzed (Participants) | 106 | 105
score on a scale
  EQ-5D 4 weeks | 0.05 [0.02 to 0.08] | 0.12 [0.08 to 0.15]
  EQ-5D 6 months: number analyzed (Participants) | 100 | 96
  EQ-5D 6 months | 0.14 [0.10 to 0.17] | 0.15 [0.12 to 0.19]
  EQ-5D 1 year: number analyzed (Participants) | 98 | 93
  EQ-5D 1 year | 0.13 [0.10 to 0.17] | 0.17 [0.14 to 0.21]

4. Other Pre Specified Outcome: Change From Baseline in Fear-Avoidance Beliefs
Description: Fear Avoidance Beliefs about physical activity and work on separate scales. The Fear avoidance about physical activity scale assesses participants' concern that physical activity will harm their back. Scores range from 0-24 with higher scores indicating greater fear of physical activity. The Fear avoidance about work scale assesses participants' concern that work-related activity will harm their back. Scores range from 0-42 with higher scores indicating greater fear of physical activity.
Time Frame: Baseline, 4 weeks, 6 months, 1 year
Population: Missing data noted across follow-up time points
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | Early Intervention
Number analyzed (Participants) | 106 | 105
units on a scale
  Fear-Avoidance Beliefs - physical activity, 4 weeks | -3.2 [-4.4 to -2.0] | -4.9 [-6.1 to -3.7]
  Fear-Avoidance Beliefs - physical activity, 6 months: number analyzed (Participants) | 100 | 96
  Fear-Avoidance Beliefs - physical activity, 6 months | -4.9 [-6.1 to -3.6] | -5.6 [-6.9 to -4.3]
  Fear-Avoidance Beliefs - physical activity, 1 year: number analyzed (Participants) | 98 | 93
  Fear-Avoidance Beliefs - physical activity, 1 year | -3.7 [-5.0 to -2.5] | -7.3 [-8.6 to -6.0]
  Fear-Avoidance Beliefs - work, 4 weeks | -1.4 [-3.1 to 0.20] | -3.0 [-4.7 to -1.3]
  Fear-Avoidance Beliefs - work, 6 months: number analyzed (Participants) | 100 | 96
  Fear-Avoidance Beliefs - work, 6 months | -3.2 [-4.9 to -1.4] | -5.0 [-6.8 to -3.3]
  Fear-Avoidance Beliefs - work, 1 year: number analyzed (Participants) | 98 | 93
  Fear-Avoidance Beliefs - work, 1 year | -2.6 [-4.3 to -0.90] | -6.2 [-8.0 to -4.4]

5. Other Pre Specified Outcome: Change From Baseline in Pain Catastrophizing Scale
Description: Self-reported measure assessing the extent to which a participant experiences catastrophizing cognitions about back pain (e.g., feelings of helplessness, hypervigilance etc.). Scores range from 13-52 with higher numbers indicating greater catastrophizing cognitions.
Time Frame: Baseline, 4 weeks, 6 months, 1 year
Population: Missing data reflected across time points
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care | Early Intervention
Number analyzed (Participants) | 106 | 105
units on a scale
  Pain catastrophizing - 4 weeks | -3.7 [-5.5 to -1.9] | -5.6 [-7.5 to -3.7]
  Pain catastrophizing - 6 months: number analyzed (Participants) | 100 | 96
  Pain catastrophizing - 6 months | -6.7 [-8.7 to -4.8] | -8.0 [-9.9 to -6.1]
  Pain catastrophizing - 1 year: number analyzed (Participants) | 98 | 93
  Pain catastrophizing - 1 year | -7.8 [-9.7 to -5.9] | -9.0 [-11.0 to -7.0]

6. Other Pre Specified Outcome: Number of Participants Utilizing Healthcare
Description: collected via online diaries
Time Frame: monthly throughout 12 month follow-up period
Population: Health care utilization over 1 year follow-up period. Participants are included in the analyses if at least one monthly utilization report was provided over the 12 month follow-up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Early Intervention
Number analyzed (Participants) | 109 | 108
Participants
  Lumbar spine surgery | 7 | 9
  Lumbar injections | 14 | 15
  Advanced Imaging | 31 | 24
  Emergency Department Visit | 11 | 10

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Usual Care | Early Intervention
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/110
Serious Adverse Events (participants affected / at risk) | 0/110 | 0/110
Other Adverse Events (participants affected / at risk) | 17/110 | 19/110
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=110) | Early Intervention (N=110)
back surgery (Musculoskeletal and connective tissue disorders) | 7 (7) | 9 (9)
injections (Musculoskeletal and connective tissue disorders) | 14 (20) | 15 (25) — Spinal injections

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-10-27): https://cdn.clinicaltrials.gov/large-docs/50/NCT02391350/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/50/NCT02391350/SAP_001.pdf